CLINICAL TRIAL: NCT05041829
Title: Dietary Sodium Intake and Blood Pressure in Living Kidney Donors: A Pilot Single-Center Crossover Single-Blind Randomized Controlled Trial
Brief Title: Dietary Sodium Intake and Blood Pressure in Living Kidney Donors
Acronym: SPLID
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Waiting for IRB approval for IRB renewal
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Ekamol Tantisattamo, MD, MPH, Associate Clinical Professor of Medicine, University of California, Irvine
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 20216478
Record Dates: First submitted 2021-09-03; First posted 2021-09-13 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Hypertension; Living Kidney Donor; Dietary Sodium Intake
Keywords: Living kidney donor; High blood pressure; Salt intake; Clinical trial
MeSH Terms: conditions — Hypertension | interventions — Sodium, Dietary

STUDY DESIGN:
Intervention Model Description: There are two 4-week experimental periods, each participant will received low and high sodium diet during one of the periods and the order of the amount of sodium diet will be determined by randomization.
Who Masked: Investigator
Masking Description: Investigator will be masked for assigned amount of dietary sodium intake of participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lowsodium (Experimental): Participants in this arm will be guided to have low dietary sodium intake of <2.3 g/day (<100 mmol/day) for 4 weeks.
  Interventions: Other: Dietary sodium
- highsodium (Active Comparator): Participants in this arm will be guided to have low dietary sodium intake of ≥4 - <6 g/day (≥174 - <261 mmo/day) for 4 weeks.
  Interventions: Other: Dietary sodium

INTERVENTIONS:
Other: Dietary sodium — Low sodium diet with sodium of <2.3 g/day (<100 mmol/day) and high sodium diet with sodium of ≥4 - <6 g/day (≥174 - <261 mmo/day)

SUMMARY:
This is a pilot study to determine the feasibility of the study design and examine the main outcome whether low dietary sodium intake is superior to high dietary sodium intake in controlling blood pressure to be within the normotensive range in living kidney donors.

DETAILED DESCRIPTION:
This is a pilot study to determine the feasibility of the study design and examine the main outcome whether low dietary sodium intake <2.3 g/day (<100 mmol/day) is superior to high dietary sodium intake ≥4 - <6 g/day (≥174 - <261 mmo/day) in controlling blood pressure (BP) to be within normotensive range, lowering systolic and diastolic blood pressures (SBP and DBP) from the baseline blood pressures, and decreasing the risk of hypertension, worsening kidney function, and proteinuria in living kidney donors between 5 and 12 months after living kidney donation?.

ELIGIBILITY:
Inclusion Criteria:

* Living kidney donors who underwent a living kidney donation at least 5 months ago but not more than 12 months
* Age ≥18 years old
* Agree to perform the procedure as per study protocol (Table 1)
* Living kidney donors with an average sitting SBP <160 mmHg at 5-month post-donation measured by automatic office blood pressure (AOBP)
* Able to sign informed consent
* Able to attend all research visits
* Woman using birth control methods other than hormonal contraception

Exclusion Criteria:

* History of previous cardiovascular (CV) events including acute MI, HF, and stroke
* Symptomatic heart failure within 5 months after living kidney donation or left ventricular ejection fraction (by any method) <35%
* CV event or procedure or hospitalization for hypertensive-related disorders within 5 months after living kidney donation
* Diagnosed with HTN or on antihypertensive medication(s) before living kidney donation
* Patients who are supposed to take BP lowering medications for reasons other than BP control but do not take those medications or take them with in appropriate doses
* Arm circumference is too small or large to allow accurate BP measurement with available 24-h ABPM machines.
* An average standing SBP ≥160 mmHg at 5-month post-donation measured by automatic office blood pressure (AOBP)
* Albuminuria that equals or is equivalent to 1 g per day by using spot urinary albumin per urine creatinine ratio (UACR) or 24-hour urinary albumin excretion rate by a 24-hour urine collection within 5 months post-donation
* Advanced kidney function defined by estimated glomerular filtration rate (eGFR) by using Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation22 of <20 ml/min/1.73m2 or requiring dialysis after living kidney donation
* Drink coffee > two 8-ounce (237 mL) cup a day or equivalence
* Drinks alcohol >3 drinks/day or >30 ml/day
* Smoking cigarette ≥10 cigarettes/day
* Take Nonsteroidal anti-inflammatory drugs (NSAIDS)
* Use hormone replacement therapy or oral contraceptives
* Pregnancy, currently trying to become pregnant
* Using birth control pills
* A medical condition likely to limit survival to less than 2 years
* Any factors that are likely to limit adherence to interventions. For example,

  * Living kidney donors who cannot come to follow up regularly per study protocol to logistically collect data from enrolled participants.
  * Active alcohol or substance abuse within the last 5 months of living kidney donation
  * Plans to move outside the clinic catchment area in the next 4 months without the ability to transfer to come to follow up at SPLID study site.
  * Significant history of poor adherences with medications or attendance at clinic visits
  * Significant concerns about participation in the study from spouse, significant other, or family members
  * Lack of support from primary health care provider
  * Residence too far from the study clinic site such that transportation is a barrier including persons who require transportation assistance provided by the SPLID clinic funds for screening or randomization visits
  * Residence in a nursing home or an assisted living
  * Clinical dementia with or without treatment with medications and cognitively unable to follow the protocol
  * Other medical, psychiatric, or behavioral factors that may interfere with study participation or the ability to follow the intervention protocol
  * Inability to obtain informed consent from participant
  * Living in the same household as an already randomized SPLID participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-11-03 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in systolic and diastolic blood pressure from baseline to post-treatment between the two treatment groups | 4 weeks after dietary intervention pre-crossover and 4 weeks after dietary intervention post-crossover
  Change in systolic and diastolic blood pressure from baseline to post-treatment between the two treatment groups, adjusting for patients' demographic and clinical differences (age, gender, BMI, and comorbidities) between the two treatment groups

SECONDARY OUTCOMES:
Hypertension | 4 weeks after dietary intervention pre-crossover and 4 weeks after dietary intervention post-crossover
  New-onset hypertension defined as systolic blood pressure >/= 130 or diastolic blood pressure >/=80 mmHg
Worsening kidney function | 4 weeks after dietary intervention pre-crossover and 4 weeks after dietary intervention post-crossover
  Increased estimated glomerular filtration rate (eGFR) >/= 25 ml/min/1.73 m2 or increased serum creatinine >/= 0.3 mg/dL
Worsening proteinuria | 4 weeks after dietary intervention pre-crossover and 4 weeks after dietary intervention post-crossover
  Increase in urinary albumin excretion rate (AER) ≥30 mg/day
Proteinuria | 4 weeks after dietary intervention pre-crossover and 4 weeks after dietary intervention post-crossover
  New-onset urinary albumin excretion rate (AER) ≥30 mg/day

CONTACTS AND LOCATIONS:
Overall Officials: Ekamol Tantisattamo, MD, MPH, Principal Investigator — University of California, Irvine
Locations (1):
- University of California Irvine Medical Center, Orange, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Result] Suthanthiran M, Strom TB. Renal transplantation. N Engl J Med. 1994 Aug 11;331(6):365-76. doi: 10.1056/NEJM199408113310606. No abstract available. PMID 7832839
- [Result] Subramanian L, Kirk R, Cuttitta T, Bryant N, Fox K, McCall M, Perry E, Swartz J, Restovic Y, Jeter A, Bernardo A, Robinson B, Perl J, Pisoni R, Perlman RL. Remote Management for Peritoneal Dialysis: A Qualitative Study of Patient, Care Partner, and Clinician Perceptions and Priorities in the United States and the United Kingdom. Kidney Med. 2019 Oct 17;1(6):354-365. doi: 10.1016/j.xkme.2019.07.014. eCollection 2019 Nov-Dec. PMID 32734216
- [Result] Davis CL, Delmonico FL. Living-donor kidney transplantation: a review of the current practices for the live donor. J Am Soc Nephrol. 2005 Jul;16(7):2098-110. doi: 10.1681/ASN.2004100824. Epub 2005 Jun 1. PMID 15930096
- [Result] Hart A, Smith JM, Skeans MA, Gustafson SK, Wilk AR, Castro S, Foutz J, Wainright JL, Snyder JJ, Kasiske BL, Israni AK. OPTN/SRTR 2018 Annual Data Report: Kidney. Am J Transplant. 2020 Jan;20 Suppl s1:20-130. doi: 10.1111/ajt.15672. PMID 31898417
- [Result] Lentine KL, Lam NN, Axelrod D, Schnitzler MA, Garg AX, Xiao H, Dzebisashvili N, Schold JD, Brennan DC, Randall H, King EA, Segev DL. Perioperative Complications After Living Kidney Donation: A National Study. Am J Transplant. 2016 Jun;16(6):1848-57. doi: 10.1111/ajt.13687. Epub 2016 Mar 10. PMID 26700551
- [Result] Lentine KL, Lam NN, Segev DL. Risks of Living Kidney Donation: Current State of Knowledge on Outcomes Important to Donors. Clin J Am Soc Nephrol. 2019 Apr 5;14(4):597-608. doi: 10.2215/CJN.11220918. Epub 2019 Mar 11. PMID 30858158
- [Result] Tantisattamo E, Dafoe DC, Reddy UG, Ichii H, Rhee CM, Streja E, Landman J, Kalantar-Zadeh K. Current Management of Patients With Acquired Solitary Kidney. Kidney Int Rep. 2019 Jul 11;4(9):1205-1218. doi: 10.1016/j.ekir.2019.07.001. eCollection 2019 Sep. PMID 31517140
- [Result] Holscher CM, Haugen CE, Jackson KR, Garonzik Wang JM, Waldram MM, Bae S, Locke JE, Reed RD, Lentine KL, Gupta G, Weir MR, Friedewald JJ, Verbesey J, Cooper M, Segev DL, Massie AB. Self-Reported Incident Hypertension and Long-Term Kidney Function in Living Kidney Donors Compared with Healthy Nondonors. Clin J Am Soc Nephrol. 2019 Oct 7;14(10):1493-1499. doi: 10.2215/CJN.04020419. Epub 2019 Sep 19. PMID 31537534
- [Result] Davis CL, Cooper M. The state of U.S. living kidney donors. Clin J Am Soc Nephrol. 2010 Oct;5(10):1873-80. doi: 10.2215/CJN.01510210. Epub 2010 Jul 15. PMID 20634322
- [Result] Boudville N, Prasad GV, Knoll G, Muirhead N, Thiessen-Philbrook H, Yang RC, Rosas-Arellano MP, Housawi A, Garg AX; Donor Nephrectomy Outcomes Research (DONOR) Network. Meta-analysis: risk for hypertension in living kidney donors. Ann Intern Med. 2006 Aug 1;145(3):185-96. doi: 10.7326/0003-4819-145-3-200608010-00006. PMID 16880460
- [Result] Lentine KL, Kasiske BL, Levey AS, Adams PL, Alberu J, Bakr MA, Gallon L, Garvey CA, Guleria S, Li PK, Segev DL, Taler SJ, Tanabe K, Wright L, Zeier MG, Cheung M, Garg AX. KDIGO Clinical Practice Guideline on the Evaluation and Care of Living Kidney Donors. Transplantation. 2017 Aug;101(8S Suppl 1):S1-S109. doi: 10.1097/TP.0000000000001769. PMID 28742762
- [Result] Svetkey LP, Sacks FM, Obarzanek E, Vollmer WM, Appel LJ, Lin PH, Karanja NM, Harsha DW, Bray GA, Aickin M, Proschan MA, Windhauser MM, Swain JF, McCarron PB, Rhodes DG, Laws RL. The DASH Diet, Sodium Intake and Blood Pressure Trial (DASH-sodium): rationale and design. DASH-Sodium Collaborative Research Group. J Am Diet Assoc. 1999 Aug;99(8 Suppl):S96-104. doi: 10.1016/s0002-8223(99)00423-x. PMID 10450301
- [Result] Gay HC, Rao SG, Vaccarino V, Ali MK. Effects of Different Dietary Interventions on Blood Pressure: Systematic Review and Meta-Analysis of Randomized Controlled Trials. Hypertension. 2016 Apr;67(4):733-9. doi: 10.1161/HYPERTENSIONAHA.115.06853. Epub 2016 Feb 22. PMID 26902492
- [Result] Yoon CY, Noh J, Lee J, Kee YK, Seo C, Lee M, Cha MU, Kim H, Park S, Yun HR, Jung SY, Jhee JH, Han SH, Yoo TH, Kang SW, Park JT. High and low sodium intakes are associated with incident chronic kidney disease in patients with normal renal function and hypertension. Kidney Int. 2018 Apr;93(4):921-931. doi: 10.1016/j.kint.2017.09.016. Epub 2017 Dec 1. PMID 29198468
- [Result] Mills KT, Chen J, Yang W, Appel LJ, Kusek JW, Alper A, Delafontaine P, Keane MG, Mohler E, Ojo A, Rahman M, Ricardo AC, Soliman EZ, Steigerwalt S, Townsend R, He J; Chronic Renal Insufficiency Cohort (CRIC) Study Investigators. Sodium Excretion and the Risk of Cardiovascular Disease in Patients With Chronic Kidney Disease. JAMA. 2016 May 24-31;315(20):2200-10. doi: 10.1001/jama.2016.4447. PMID 27218629
- [Result] Anjum S, Muzaale AD, Massie AB, Bae S, Luo X, Grams ME, Lentine KL, Garg AX, Segev DL. Patterns of End-Stage Renal Disease Caused by Diabetes, Hypertension, and Glomerulonephritis in Live Kidney Donors. Am J Transplant. 2016 Dec;16(12):3540-3547. doi: 10.1111/ajt.13917. Epub 2016 Jul 12. PMID 27287605
- [Result] Lee JH, Kim SC, Han DJ, Chang JW, Yang WS, Park SK, Lee SK, Park JS, Kim SB. Risk factors for MDRD-GFR of less than 60 mL/min per 1.73 m2 in former kidney donors. Nephrology (Carlton). 2007 Dec;12(6):600-6. doi: 10.1111/j.1440-1797.2007.00852.x. PMID 17995588
- [Result] Mjoen G, Hallan S, Hartmann A, Foss A, Midtvedt K, Oyen O, Reisaeter A, Pfeffer P, Jenssen T, Leivestad T, Line PD, Ovrehus M, Dale DO, Pihlstrom H, Holme I, Dekker FW, Holdaas H. Long-term risks for kidney donors. Kidney Int. 2014 Jul;86(1):162-7. doi: 10.1038/ki.2013.460. Epub 2013 Nov 27. PMID 24284516
- [Result] Young A, Storsley L, Garg AX, Treleaven D, Nguan CY, Cuerden MS, Karpinski M. Health outcomes for living kidney donors with isolated medical abnormalities: a systematic review. Am J Transplant. 2008 Sep;8(9):1878-90. doi: 10.1111/j.1600-6143.2008.02339.x. Epub 2008 Jul 28. PMID 18671676
- [Result] Sacks FM, Svetkey LP, Vollmer WM, Appel LJ, Bray GA, Harsha D, Obarzanek E, Conlin PR, Miller ER 3rd, Simons-Morton DG, Karanja N, Lin PH; DASH-Sodium Collaborative Research Group. Effects on blood pressure of reduced dietary sodium and the Dietary Approaches to Stop Hypertension (DASH) diet. DASH-Sodium Collaborative Research Group. N Engl J Med. 2001 Jan 4;344(1):3-10. doi: 10.1056/NEJM200101043440101. PMID 11136953
- [Result] Levey AS, Stevens LA, Schmid CH, Zhang YL, Castro AF 3rd, Feldman HI, Kusek JW, Eggers P, Van Lente F, Greene T, Coresh J; CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration). A new equation to estimate glomerular filtration rate. Ann Intern Med. 2009 May 5;150(9):604-12. doi: 10.7326/0003-4819-150-9-200905050-00006. PMID 19414839
- [Result] Institute of Medicine (US) Committee to Review Dietary Reference Intakes for Vitamin D and Calcium; Ross AC, Taylor CL, Yaktine AL, Del Valle HB, editors. Dietary Reference Intakes for Calcium and Vitamin D. Washington (DC): National Academies Press (US); 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK56070/ PMID 21796828
- [Result] Low PA, Opfer-Gehrking TL, McPhee BR, Fealey RD, Benarroch EE, Willner CL, Suarez GA, Proper CJ, Felten JA, Huck CA, et al. Prospective evaluation of clinical characteristics of orthostatic hypotension. Mayo Clin Proc. 1995 Jul;70(7):617-22. doi: 10.4065/70.7.617. PMID 7791382
- [Result] Pickering TG, Hall JE, Appel LJ, Falkner BE, Graves J, Hill MN, Jones DW, Kurtz T, Sheps SG, Roccella EJ; Subcommittee of Professional and Public Education of the American Heart Association Council on High Blood Pressure Research. Recommendations for blood pressure measurement in humans and experimental animals: Part 1: blood pressure measurement in humans: a statement for professionals from the Subcommittee of Professional and Public Education of the American Heart Association Council on High Blood Pressure Research. Hypertension. 2005 Jan;45(1):142-61. doi: 10.1161/01.HYP.0000150859.47929.8e. Epub 2004 Dec 20. PMID 15611362
- [Result] Cox DR. Regression models and life tables (with discussion). Journal of the Royal Statistical Society, Series B 34, 187-220, 1972.